CLINICAL TRIAL: NCT04906083
Title: The Efficacy and Safety of Avatrombopag in Patients With End-stage Liver Disease and Thrombocytopenia: A Multicenter, Prospective, Randomized Controlled Trial（EAST）
Brief Title: Avatrombopag in Patients With End-stage Liver Disease and Thrombocytopenia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Anhui Provincial Hospital (Other Government); The First Affiliated Hospital of Nanchang University (Other); Taihe Hospital, Hubei University of Medicine (Unknown); The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Qin Ning, Director of Department of Infectious Diseases, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJ20210517
Record Dates: First submitted 2021-05-17; First posted 2021-05-28 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Liver Failure; Thrombocytopenia; Decompensated Cirrhosis
Keywords: end-stage liver disease; thrombocytopenia; avatrombopag; efficacy; safety
MeSH Terms: conditions — Liver Failure; Thrombocytopenia; End Stage Liver Disease | interventions — avatrombopag; Glutathione; Hepatocyte Growth Factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Avatrombopag+Standard medical treatment
  Interventions: Drug: Avatrombopag; Drug: Standard medical treatment
- Control group (Other): Standard medical treatment
  Interventions: Drug: Standard medical treatment

INTERVENTIONS:
Drug: Avatrombopag — Avatrombopag:
  PLT：30~50×10^9/L patients, 40 mg/d; PLT：<30×10^9/L patients, 60 mg/d.
  Arms: Intervention group
Drug: Standard medical treatment — Standard medical treatment included transmetil, compound glycyrrhizinate, reduced glutathione and hepatocyte growth factor, et. al.
  Other Names: transmetil, compound glycyrrhizinate, reduced glutathione and hepatocyte growth factor, et. al.

SUMMARY:
End stage liver disease is prone to thrombocytopenia. This study is a multi-center, randomized, prospective, randomized controlled Phase IV Clinical trial to discuss the Efficacy and Safety of Avatrombopag in Patients with End-stage Liver Disease and Thrombocytopenia.

DETAILED DESCRIPTION:
End stage liver disease is prone to thrombocytopenia. This study aims to discuss the Efficacy and Safety of Avatrombopag in Patients with End-stage Liver Disease and Thrombocytopenia in a multicenter, prospective, randomized controlled trial. The patients were divided into one of the groups according to if receiving avatrombopag. Avatrombopag was taken to maintain platelet count 50~100×10^9/L. Starting dose is recommended according to the patient's baseline platelet count level. Routine treatment was taken in the Control group and Interventional group. This trial will take about 2 to 2.5 years from the first participant signing an informed consent form (ICF) until all study-related telephone follow-ups or visits end.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women greater than or equal to 18 years of age;
2. Baseline platelet count <50×10^9/L;
3. End-stage liver disease, including acute-on-chronic liver failure, acute decompensation of liver cirrhosis, chronic liver failure;
4. Women of childbearing potential must agree to use a highly effective method of contraception from the beginning of Baseline Visit until the end of treatment (includes implantable contraception, injectable contraception, hormonal combination contraception [including vaginal rings], intra-uterine devices or vasectomy). The barrier contraception with or without spermicide alone, double barrier contraception and oral contraceptives are inadequate;
5. Subject is able to understand the study and willing to follow the protocol and sign informed consent voluntarily before Baseline Visit;
6. Subject meet the criteria according to the opinion of the researchers.

Exclusion Criteria:

1. Subject has a history of arterial or venous thrombosis within the previous 6 months of baseline;
2. Known portal vein blood flow velocity rate <10 cm/second or previous occurrence of a portal vein thrombosis within 6 months of Baseline;
3. Known any history of primary blood (e.g, immune thrombocytopenia, myelodysplastic syndrome, aplastic anemia);
4. Subject has a known medical history of genetic prothrombotic syndromes (e.g, Factor V Leiden prothrombin G20210A, antithrombin III (AT III) deficiency);
5. Subject has a recent history (within the previous 6 months) of significant cardiovascular diseases (e.g., exacerbation of congestive heart failure, arrhythmias known to increase the risk of thromboembolic events [e.g. atrial fibrillation], coronary or peripheral artery stent placement or angioplasty, and coronary or peripheral artery bypass grafting);
6. Female subjects who are lactating or pregnant at the Baseline Visit (as documented by a positive serum beta-human chorionic gonadotropin [β-hCG] test with a minimum sensitivity of 25 IU/L or equivalent units of β-hCG) or are planning to become pregnant during the study;
7. The subject has a hypersensitivity to Avatrombopag or any of its excipients;
8. Subjects with drug-induced thrombocytopenia;
9. Subjects whose Life expectation ≤6 months;
10. Subject with a current malignancy;
11. Subjects with HIV infection;
12. At screening, active infection was not effectively controlled by systemic antibiotic therapy;
13. The Investigator believe that any accompanying medical history may affect the safety of the subjects to complete the study;
14. The Investigator believe that there are any other factors that are not suitable for inclusion or affect participation or completion of the study;
15. Subject is enrolled in another clinical study with any investigational drug or device within previous 30 days of the Baseline Visit, but are allowed to participate in observational studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Platelet count response time | 24 weeks
  Platelet count response time(PLT) refers to condition of PLT during 24 weeks between the Intervention group and Control group.

SECONDARY OUTCOMES:
Adverse Event (thrombotic events, bleeding events, etc.) incidence; | 24 weeks
  Adverse Event refers to the incidence rate of adverse event between the two groups during 24 weeks
Incidence of complications of liver cirrhosis (infection, etc.) | 24 weeks
  Incidence of complications of liver cirrhosis refers to the incidence rate of complications between the two groups during 24 weeks
Patients without platelet transfusion or rescue due to bleeding | 24 weeks
  Patients without platelet transfusion or rescue due to bleeding refers to the patients rate without platelet transfusion or rescue due to bleeding between the two groups at 24 week
Proportion of patients readmitted | 24 weeks
  Proportion of patients readmitted refers to the readmission rate within 24 weeks between the Intervention group and Control group
Changes in total bilirubin level | 24 weeks
  Changes in total bilirubin level refers to the changes of total bilirubin at 24 week compared to baseline between the Intervention group and Control group.
Changes in alanine aminotransferase level | 24 weeks
  Changes in alanine aminotransferase level refers to the changes of alanine aminotransferase at 24 week compared to baseline between the Intervention group and Control group.
Changes in albumin level | 24 weeks
  Changes in albumin level refers to the changes of albumin at 24 week compared to baseline between the Intervention group and Control group.
Changes in prothrombin time level | 24 weeks
  Changes in prothrombin time level refers to the changes of prothrombin time at 24 week compared to baseline between the Intervention group and Control group.
Changes in international normalized ratio level | 24 weeks
  Changes in international normalized ratio level refers to the changes of international normalized ratio at 24 week compared to baseline between the Intervention group and Control group.

CONTACTS AND LOCATIONS:
Overall Officials: Qin Ning, MD., PhD., Study Chair — Department of Infectious Disease, Tongji Hospital, Tongji Medical College, HUST
Locations (1):
- Department of infectious disease, Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided